CLINICAL TRIAL: NCT03962790
Title: Clinical Evaluation of Etafilcon A Contact Lenses Using a Novel Manufacturing Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR-6324
Record Dates: First submitted 2019-05-23; First posted 2019-05-24 (Actual); Results first posted 2020-08-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Visual Acuity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Test/Control (Experimental): Eligible subjects that are habitual wearers of hydrogel daily disposable contact lenses in both eyes will be randomly assigned to one of two sequences, (Test/Control) or (Control/Test).
  Interventions: Device: 1-DAY ACUVUE® MOIST
- Control/Test (Experimental): Eligible subjects that are habitual wearers of hydrogel daily disposable contact lenses in both eyes will be randomly assigned to one of two sequences, (Test/Control) or (Control/Test).
  Interventions: Device: 1-DAY ACUVUE® MOIST

INTERVENTIONS:
Device: 1-DAY ACUVUE® MOIST — etafilcon A contact lenses made with a new manufacturing technology
  Other Names: Test
Device: 1-DAY ACUVUE® MOIST — etafilcon A contact lenses made with the current manufacturing technology
  Other Names: Control

SUMMARY:
This study is a multi-site, randomized, double-masked, 2×2 crossover design, 1-week dispensing study. Subjects will wear both Test and Control lenses in each eye in a random order for 1-week each as a daily disposable modality with a wash-out period of 1 week between the wearing periods.

ELIGIBILITY:
Inclusion Criteria:

* Potential subjects must satisfy all of the following criteria to be enrolled in the study:

  1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
  2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
  3. Must be at least 18 and not more than 70 years of age (including 70) at the time of screening.
  4. The subject must be a habitual and adapted wearer of hydrogel daily disposable brand contact lenses in both eyes (at least 1 month of daily wear).
  5. The subject must have normal eyes (i.e., no ocular medications or infections of any type).
  6. The subject's required spherical contact lens prescription must be in the range of -0.50 to -6.00 D in each eye.
  7. The subject's refractive cylinder must be < 0.75D in each eye.
  8. The subject must have best corrected visual acuity of 20/25 or better in each eye.

     Exclusion Criteria:
* Potential subjects who meet any of the following criteria will be excluded from participating in the study:

  1. Currently pregnant or lactating (subjects who become pregnant during the study will be discontinued).
  2. Any systemic disease, autoimmune disease, or use of medication that may interfere with contact lens wear.
  3. Any previous, or planned, ocular or interocular surgery (e.g., radial keratotomy, PRK, LASIK, etc.).
  4. Any ocular infection.
  5. Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.
  6. Monovision or multi-focal contact lens correction.
  7. Participation in any contact lens or lens care product clinical trial within 14 days prior to study enrollment.
  8. History of binocular vision abnormality or strabismus.
  9. Any infectious disease (e.g., hepatitis, tuberculosis) or a contagious immunosuppressive disease (e.g., HIV, by self-report).
  10. Suspicion of or recent history of alcohol or substance abuse.
  11. History of serious mental illness.
  12. History of seizures.
  13. Employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician)
  14. Any ocular allergies, infections or other ocular abnormalities that are known to interfere with contact lens wear and/or participation in the study. This may include, but not be limited to entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, or corneal distortion
  15. Any Grade 3 or greater slit lamp findings (e.g., edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) on the Food and Drug Administration (FDA) classification scale
  16. Any previous history or signs of a contact lens-related corneal inflammatory event (e.g., past peripheral ulcer or round peripheral scar), or any other ocular abnormality that may contraindicate contact lens wear.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2019-07-10 (Actual); Study Completion 2019-07-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Maitland Vision Center, Maitland, Florida
  - Eyecare Associates, LLP, Bloomington, Illinois
  - Manhattan Vision Associates, New York, New York
  - Sacco Eye Group, Vestal, New York
  - Eyecare Professionals of Powell, Powell, Ohio
  - Frazier Vision, Tyler, Texas

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 95 participants were enrolled in this study however one participant was never randomized due to screen failure therefore, 94 participants were randomized to receive study drug.
Groups:
- Test/Control: Subjects randomized to this sequence received the Test lens during the first period and then received the control lens during the second period.
- Control/Test: Subjects randomized to this sequence received the Control lens during the first period and then received the Test lens during the second period.
Period: Period 1
Arm/Group | Test/Control | Control/Test
Started | 48 | 46
Completed | 45 | 44
Not Completed | 3 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Failed to meet all eligibility criteria | 1 | 1
Not completed — No Longer Meets Eligibility Criteria | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Period 2
Arm/Group | Test/Control | Control/Test
Started | 45 | 44
Completed | 45 | 44
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Set: All subjects dispensed a study lens.
Arm/Group | Overall Set
Number analyzed (Participants) | 94
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.7 (9.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64
  Male | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 78
  More than one race | 6
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Comfort Score
Description: Overall comfort score was assessed using the Contact Lens User Experience (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (standard deviation [SD] 20), where higher scores indicate a more favorable/positive response. A 5-point increase in an average CLUE score translates into 10% shift in the distribution of scores for the population of soft disposable contact lens wearers.
Time Frame: 1-Week Follow-up
Population: All subjects who had successfully completed all visits and did not substantially deviate from the protocol.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Etafilcon A Test for Novel: Subjects who wore the Test lens made with a novel manufacturing technology in either the first or second period of the study.
- Etafilcon A Control for Current: Subjects that wore the Control lens made with the current manufacturing technology in either the first or second period of the study.
Arm/Group | Etafilcon A Test for Novel | Etafilcon A Control for Current
Number analyzed (Participants) | 89 | 89
Units on a scale | 56.52 (20.631) | 55.72 (22.567)
Statistical Analysis 1: Comparison: Etafilcon A Test for Novel vs Etafilcon A Control for Current; Bayesian repeated measurement random-effects model was used to compare between Test and Control lenses; Test type: Non-Inferiority — Non-inferiority was declared if the lower bound of the credible interval (CrI) of the mean difference between Test and Control was greater than -5; Posterior Mean Difference = 0.09, 95% CI 2-sided [-4.37 to 4.65], Standard Deviation 2.281 — Posterior mean difference was calculated as Test - Control

2. Primary Outcome: Overall Vision Score
Description: Overall quality of vision was assessed using the Contact Lens User Experience (CLUE) questionnaire. CLUE is a validated patient reported outcomes (PRO) questionnaire to assess patient-experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response. A 5-point increase in an average CLUE score translates into 10% shift in the distribution of scores for the population of soft disposable contact lens wearers.
Time Frame: 1-Week Follow-up
Population: All subjects who had successfully completed all visits and did not substantially deviate from the protocol.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etafilcon A Test for Novel | Etafilcon A Control for Current
Number analyzed (Participants) | 89 | 89
Units on a scale | 61.65 (19.161) | 62.47 (20.670)
Statistical Analysis 1: Comparison: Etafilcon A Test for Novel vs Etafilcon A Control for Current; Bayesian repeated measurement random-effects model was used to compare between Test and Control lenses; Test type: Non-Inferiority — Non-inferiority is established if the lower limit of the 95% credible interval is above -5 points in CLUE Scale; Posterior Mean Difference = -1.02, 95% CI 2-sided [-4.07 to 2.06], Standard Deviation 1.565 — Posterior mean difference was calculated as Test - Control

3. Secondary Outcome: LogMAR Visual Performance Scale
Description: Visual acuity measured via Early Treatment Diabetic Retinopathy Study (ETDRS) charts (logMAR) can take on any possible value. A value of 0.0 logMAR equates to 20/20 vision on a Snellen Scale. Lower values indicate better visual performance. The average visual performance is reported for each lens type on high contrast dim light and low contrast bright light.
Time Frame: 1-Week follow-up
Population: All subjects who had successfully completed all visits and did not substantially deviate from the protocol.
Measure: Mean (Standard Deviation); unit: logMAR units
Units Other Than Participants: Eyes
Arm/Group | Etafilcon A Test for Novel | Etafilcon A Control for Current
Number analyzed (Participants) | 89 | 89
Number analyzed (Eyes) | 178 | 178
logMAR units
  High Contrast Dim | -0.018 (0.1276) | -0.017 (0.1173)
  Low Contrast Bright | 0.022 (0.0915) | 0.024 (0.0924)
Statistical Analysis 1: Comparison: Etafilcon A Test for Novel vs Etafilcon A Control for Current; Bayesian repeated measurement random-effects model was used to compare between Test and Control lenses; Test type: Non-Inferiority — Non-inferiority was declared if the upper bound of the CrI of the mean difference between Test and Control was less than 0.05; Posterior Mean Difference = -0.001, 95% CI 2-sided [-0.012 to 0.010], Standard Deviation 0.0054 — Posterior mean difference was calculated as Test - Control
Statistical Analysis 2: Comparison: Etafilcon A Test for Novel vs Etafilcon A Control for Current; Bayesian repeated measurement random-effects model was used to compare between Test and Control lenses; Test type: Non-Inferiority — [test comment as in outcome 3, analysis 1]; Posterior Mean Difference = -0.002, 95% CI 2-sided [-0.014 to 0.009], Standard Deviation 0.0057 — Posterior mean difference was calculated as Test - Control

4. Secondary Outcome: Average Daily Wear Time
Description: Average daily wear time was calculated as the number of hours between participants reported time of insertion and time of removal of the study lenses, on an average day, at 1-Week follow-up evaluation.
Time Frame: 1-Week follow-up
Population: All subjects who had successfully completed all visits and did not substantially deviate from the protocol.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Etafilcon A Test for Novel | Etafilcon A Control for Current
Number analyzed (Participants) | 89 | 89
Hours | 14.22 (1.937) | 14.16 (1.866)
Statistical Analysis 1: Comparison: Etafilcon A Test for Novel vs Etafilcon A Control for Current; Bayesian repeated measurement random-effects model was used to compare between Test and Control lenses; Test type: Non-Inferiority — Non-inferiority was declared if the lower bound of the CrI of the mean difference between Test and Control was greater than -1; Posterior Mean Difference = 0.02, 95% CI 2-sided [-0.32 to 0.34], Standard Deviation 0.168 — Posterior mean difference was calculated as Test - Control

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study. Approximately 3-4 Weeks per participant
Description: All participants dispensed at least 1 study lens.
Arm/Group | Etafilcon A Test for Novel | Etafilcon A Control for Current
All-Cause Mortality (participants affected / at risk) | 0/92 | 0/91
Serious Adverse Events (participants affected / at risk) | 0/93 | 0/90
Other Adverse Events (participants affected / at risk) | 0/93 | 0/90

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-26): https://cdn.clinicaltrials.gov/large-docs/90/NCT03962790/Prot_SAP_000.pdf